CLINICAL TRIAL: NCT01039935
Title: Genetic Basis of Odor Discrimination
Status: Completed | Type: Observational
Sponsor: Rockefeller University (Other)
Responsible Party: Sponsor
Other Study IDs: LVO-0684
Record Dates: First submitted 2009-12-23; First posted 2009-12-25 (Estimated); Last update posted 2012-09-06 (Estimated); Status verified 2012-09

CONDITIONS: Non-smokers
Keywords: Odor Discrimination

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample taken
Oversight: Data Monitoring Committee: No

SUMMARY:
Prior to the main study we will perform a pilot study on 60 subjects. The purpose of the pilot study is to identify the range of odor concentrations that will be used in the main study and to optimize the tasks performed in the main study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-50
2. Current non-smokers

Exclusion Criteria:

1. Current smokers
2. Allergy to fragrances or smells of any kind
3. Active head cold, upper respiratory infection, or seasonal nasal allergies
4. History of nasal health problems, including endoscopic nasal surgery for sinus conditions or polyp removal.
5. Pre-existing medical condition that has caused anosmia or near total loss of the sense of smell, such as: head injury, cancer therapy, radiation to head and neck, or alcoholism

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers
Sampling Method: Probability Sample
Enrollment: 512 (Actual)
Dates: Start 2009-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Percentage of correct responses when discriminating between (-)-carvone and (+)-carvone, isovaleric acid and isobutyric acid, androstenone and androstadienone DNA sequence of ORs sensitive to these odors | 3 years

SECONDARY OUTCOMES:
concentration at which odors need to be added to allow for discrimination; thresholds to all six odors; verbal descriptors assigned to all six odors | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Vosshall, PhD, Principal Investigator — The Rockefeller University
Locations (1):
- The Rockefeller University, New York, New York, United States